CLINICAL TRIAL: NCT00688025
Title: Magnetoencephalographic Localization of Ramelteon's Effects on Brain Function and Cortical Arousal in Insomnia
Brief Title: Magnetoencephalographic (MEG) Localization of Ramelteon's Effects on Brain Function and Cortical Arousal in Insomnia
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Christopher Drake, Ph.D., Henry Ford Health System
Other Study IDs: 07-033R
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Insomniacs: Individuals reporting difficulty falling asleep or staying asleep within the past month for more than 3 days per week. Individuals much also meet screening criteria based on an overnight polysomnograph of latency to persistent sleep >20 minutes and/or >60 minutes of wake after sleep onset.
- 2: Controls: Individuals reporting no difficulty falling asleep or staying asleep and objective sleep measures based on an overnight polysomnograph of latency to persistent sleep <20 minutes and/or <60 minutes of wake after sleep onset.

SUMMARY:
The present protocol will utilize simultaneous recording of brain activity during attention and memory tasks in insomnia participants after ramelteon vs. zolpidem vs. placebo administration. The investigators hypothesize that amplitudes of associated with memory will be unchanged by ramelteon, whereas zolpidem will significantly reduce brain activity associated with stimulus processing as evidenced by abnormal reduction in the amplitude of specific brain regions relative to placebo.

DETAILED DESCRIPTION:
The proposed research has two specific aims: 1) demonstrate that ramelteon has no effect on event related potential components that reflect basic sensory processes (P1 and N1), and will not impair attention and memory processes, whereas the benzodiazepine receptor agonist zolpidem will significantly reduce (relative to placebo) the amplitude of these event related potential components throughout the cerebral cortex and 2) show that ramelteon reduces the abnormal hyperarousal in insomnia as reflected through a reduction in the contingent negative variation component of the event related potential across frontal and parietal brain regions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with no secondary condition to insomnia.

Exclusion Criteria:

* Healthy individuals with no insomnia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Insomniacs, individuals with difficulty falling asleep or staying asleep.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Drake, Ph.D., Principal Investigator — Henry Ford Hospital Sleep Disorders & Research Center
Locations (1):
- Henry Ford Hospital Sleep Disorders & Research Center, Detroit, Michigan, United States